CLINICAL TRIAL: NCT01303796
Title: A Phase III Randomized Study of Oral Sapacitabine in Elderly Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: A Study of Oral Sapacitabine in Elderly Patients With Newly Diagnosed Acute Myeloid Leukemia
Acronym: SEAMLESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYC682-12
Record Dates: First submitted 2011-02-21; First posted 2011-02-25 (Estimated); Results first posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — sapacitabine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sapacitabine-decitabine alternating (Experimental): Arm A sapacitabine administered in alternating cycles with decitabine
  Interventions: Drug: Sapacitabine; Drug: Decitabine
- Decitabine (Active Comparator): Arm C Decitabine
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Sapacitabine — Oral sapacitabine capsules
  Other Names: CYC682
  Arms: Sapacitabine-decitabine alternating
Drug: Decitabine — Decitabine intravenous
  Other Names: Decitabine intravenous

SUMMARY:
This Phase 3 study assesses two drug regimens as the initial treatment of patients who are at least 70 years of age and have newly diagnosed acute myeloid leukemia (AML) for whom the doctor does not recommend the use of standard intensive treatment or the patient has decided not to receive standard intensive treatment after being fully informed about its benefits and risks by his/her doctor. The two drug regimens are sapacitabine administered in alternating cycles with decitabine or decitabine alone. The purpose of the study is to learn which drug regimen is more likely to keep AML in check as long as possible.

DETAILED DESCRIPTION:
This is a multicenter, randomized, Phase 3 study ("SEAMLESS") comparing two drug regimens (arms) as the front-line treatment of elderly patients aged 70 years or older with newly diagnosed acute myeloid leukemia (AML) who are not candidates for intensive induction chemotherapy. In Arm A, sapacitabine is administered in alternating cycles with decitabine, and in Arm C decitabine is administered alone. The primary efficacy endpoint is overall survival. The study is designed to demonstrate an improvement in overall survival of Arm A versus Arm C.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML based on WHO (World Health Organization) classification
* Age 70 years or older for whom the treatment of choice is low-intensity therapy by investigator assessment or who has refused intensive induction therapy recommended by investigator
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* Adequate renal function
* Adequate liver function
* Able to swallow capsules
* Agree to practice effective contraception
* Ability to understand and willingness to sign the informed consent form

Exclusion Criteria:

* AML is of the sub-type of acute promyelocytic leukemia or extramedullary myeloid tumor without bone marrow involvement
* Having received any systemic anti-cancer therapy for AML or received treatment with hypomethylating agents or cytotoxic chemotherapy for preceding myelodysplastic syndrome (MDS) or myeloproliferative disease (MPD)
* Known or suspected central nervous system (CNS) involvement by leukemia
* Uncontrolled intercurrent illness
* Known hypersensitivity to decitabine
* Known to be HIV-positive

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 482 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop M Kantarjian, M.D., Study Chair — M.D. Anderson Cancer Center
Locations (118):
- United States (39):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Scripps Cancer Center, La Jolla, California
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - Norwalk Hospital, Norwalk, Connecticut
  - Shands Cancer Hospital at University of Florida, Gainesville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - St. Francis Medical Group Oncology and Hematology Specialists, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Maryland Greenbaum Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - St. Louis University Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth - Hitchcock Medical Center, Lebanon, New Hampshire
  - John Theurer Cancer Center at the Hackensack University Medical Center, Hackensack, New Jersey
  - Westchester Hematology Oncology Group, PC, Hawthorne, New York
  - Beth Israel Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Saint Francis Hospital, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- Austria (7):
  - Medizinische Universitaetsklinik, Innsbruck
  - Elisabethinen Krankenhaus, Linz
  - Krankenhaus der Barmherzigen Schwestern, Linz
  - Univ. Klinik fur Innere Medizin III LKH, Salzburg
  - AKH Wien, Vienna
  - Hanusch Krankenhaus, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (5):
  - Ziekenhuis Netwerk Antwerpen Stuivenberg, Antwerp
  - AZ Sint-Jan Brugge-Oostende, Bruges
  - Universite Catholique de Louvain, Brussels
  - Centre Hospitalier De Jolimont-Lobbes, La Louvière
  - Cliniques Universitaires UCL de Mont-Godinne, Yvoir
- France (13):
  - CHU d'Amiens Hopital Sud, Amiens
  - Centre Hospitalier de la Cote Basque, Bayonne
  - CHU de Lyon - Hopital Edouard Herriot, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHRU De Montpellier Hopital St. Eloi, Montpellier
  - Centre Hospitalier De Mulhouse, Mulhouse
  - Hopital St Louis Universite Paris 7, Paris
  - Centre Hospitalier de Perigueux, Périgueux
  - Centre Hospitalier d'Annecy, Pringy
  - Centre Hospitalier de Saint-Brieuc Yves Ie Foll, Saint-Brieuc
  - CHU de Strasbourg - Hopital Civil, Strasbourg
  - Strasbourg Oncologie Liberale, Strasbourg
  - CHU de Tours Hopital Bretonneau, Tours
- Germany (11):
  - Universitaetsklinikum Charite Berlin, Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Carl-Gustav-Carus Dresden, Dresden
  - St. Johannes Hospital, Duisburg
  - Klinikum Frankfurt Hoechst, Frankfurt
  - Asklepios Klinik Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - SLK Kliniken Heilbronn, Heilbronn
  - Klinikum St. Georg, Leipzig
  - Johannes Wesling Klinikum, Minden
  - TU Muenchen, München
  - Universitaetsklinikum Muenster, Münster
- Hungary (3):
  - University of Debrecen, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Kaposi Mor Oktato Korhaz, Kaposvár
- Italy (15):
  - AOU Ospedali Riuniti Umberto I, Ancona
  - AO Ospedali Riuniti di Bergamo, Bergamo
  - Universita di Bologna Ist Ematologia Oncologia Medica Seragnoli, Bologna
  - AO Spedali Civili di Brescia, Brescia
  - Universita Cattolica del Sacro Cuore, Campobasso
  - AOU Careggi, Florence
  - AOU San Martino IST, Genova
  - PO Vito Fazzi, Lecce
  - Ospedale San Raffaele, Milan
  - AORN Antonio Cardarelli, Napoli
  - Uni. Napoli Ospedale Federico lI, Napoli
  - AOU Maggiore della Carità di Novara, Novara
  - AOOR Villa Sofia Cervello di Palermo, Palermo
  - Policlinico San Matteo Di Pavia, Pavia
  - AOU San Luigi Gonzaga, Torino
- Poland (6):
  - Akademickie Centrum Kliniczne Szpital Akademii Medycznej w Gdansku, Gdansk
  - Wojewodzki Szpital Specjalistyczny, Legnica
  - Wojewódzki Szpital Specjalistyczny w Legnicy, Legnica
  - University of Lodz N. Copernicus Memorial Hospital, Lodz
  - IHT Instytut Hematologii I Transfuzjologii w Warszawie, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Wroclawiu, Wroclaw
- Spain (15):
  - Hospital Universitari Germans Trias i Pujol ICO Badalona, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital De La Santa Creu Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Clínica Universidad de Navarra, Pamplona
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Clinico Universitario, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari "La Fe", Valencia
- Sweden (2):
  - Sunderby Hospital, Luleå
  - Skåne Universitetssjukhus Univ Hospital Lund, Lund
- Inselspital Bern, Bern, Switzerland
- Kings College Hospital and Guys and St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kantarjian HM, Begna KH, Altman JK, Goldberg SL, Sekeres MA, Strickland SA, Arellano ML, Claxton DF, Baer MR, Gautier M, Berman E, Seiter K, Solomon SR, Schiller GJ, Luger SM, Butrym A, Gaidano G, Thomas XG, Montesinos P, Rizzieri DA, Quick DP, Venugopal P, Gaur R, Maness LJ, Kadia TM, Ravandi F, Buyse ME, Chiao JH. Results of a randomized phase 3 study of oral sapacitabine in elderly patients with newly diagnosed acute myeloid leukemia (SEAMLESS). Cancer. 2021 Dec 1;127(23):4421-4431. doi: 10.1002/cncr.33828. Epub 2021 Aug 23. PMID 34424530
- See also: Results of a randomized phase 3 study of oral sapacitabine in elderly patients with newly diagnosed acute myeloid leukemia (SEAMLESS) — https://pubmed.ncbi.nlm.nih.gov/34424530/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study comprised a single-arm Lead-in phase to confirm the safety and tolerability of administering sapacitabine in alternating cycles with decitabine prior to patients being enrolled in the parallel group, randomized Phase III phase to compare the two treatment arms. 21 patients were enrolled in the Lead-in phase.
Groups:
- Lead In Phase: Decitabine alternating with sapacitabine (n=21). Patients followed for safety. Lead in group is not included in ITT analysis of randomized portion of the trial.
- Sapacitabine-decitabine Alternating: Arm A patients received sapacitabine capsules in alternating cycles with decitabine i.e., Cycle 1=decitabine, Cycle 2=sapacitabine, Cycle 3=decitabine, Cycle 4=sapacitabine, etc. Arm A is preceded by a Lead-in phase in selected patients.
  Sapacitabine: Oral capsules; 300 mg twice daily (b.i.d.) orally x 3 consecutive days/week x 2 weeks every 8 weeks Decitabine: Decitabine intravenous; 20 mg/m2 infused over 1 hour intravenously/day x 5 consecutive days every 8 weeks Patients continued treatment until one of the following occurred: clinically significant progressive disease; lack of efficacy; unacceptable toxicity; patient withdrawal of consent; investigator's assessment; intercurrent illness or changes in patient's condition that rendered the patient ineligible or continuing treatment unsafe, or regular follow-up impossible; a pattern of non-compliance with study medication or protocol-required evaluations and follow-up; or termination of the clinical trial by the sponsor.
- Decitabine: Arm C patients received decitabine infusion.
  Decitabine: Intravenous; 20 mg/m2 infused over 1 hour intravenously/day x 5 consecutive days every 8 weeks
  Patients continued treatment until one of the following occurred: clinically significant progressive disease; lack of efficacy; unacceptable toxicity; patient withdrawal of consent; investigator's assessment that it was in the best interest of the patient to withdraw; intercurrent illness or changes in patient's condition that rendered the patient ineligible or continuing treatment unsafe, or regular follow-up impossible; a pattern of non-compliance with study medication or protocol-required evaluations and follow-up; or termination of the clinical trial by the sponsor.
Period: Lead In Phase
Arm/Group | Lead In Phase | Sapacitabine-decitabine Alternating | Decitabine
Started | 21 | 0 (Intend-to-Treat study subject population) | 0 (Intend-to-Treat study subject population)
Completed | 21 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Randomized Phase III
Arm/Group | Lead In Phase | Sapacitabine-decitabine Alternating | Decitabine
Started | 0 | 241 | 241
Completed | 0 | 241 | 241
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Elderly patients with newly diagnosed acute myeloid leukemia (AML) for whom the treatment of choice was low-intensity therapy by investigator assessment, or who had refused intensive induction therapy recommended by the investigator.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine | Total
Number analyzed (Participants) | 241 | 241 | 482
Age, Continuous [Median (Full Range); unit: years] | 78 [70 to 92] | 77 [70 to 92] | 77 [70 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 95 | 197
  Male | 139 | 146 | 285
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 212 | 194 | 406
  Black | 6 | 17 | 23
  Asian or Pacific Islander | 1 | 3 | 4
  Hispanic | 6 | 3 | 9
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 2 | 3 | 5
  Unknown | 13 | 21 | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The distribution of overall survival was estimated by the method of Kaplan and Meier. A log-rank analysis stratified by randomization stratification factors was used to compare overall survival between Arm A (decitabine/sapacitabine) versus Arm C (decitabine). Cox proportional hazards models were used to identify predictive factors for overall survival.
Time Frame: up to 43 months
Population: Patients >= 70 years with histologically or pathologically confirmed AML; not treated by systemic therapy; on low-intensity therapy by investigator assessment or the patient has refused standard induction chemotherapy; no prior treatment with HMA or other anti-cancer agents; ECOG status 0-2; adequate hepatic and renal function
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 226 | 218
Months | 5.9 [4.7 to 8.0] | 5.7 [4.9 to 8.2]
Statistical Analysis 1: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; The phase III part planned to randomize 485 patients, about 243 per arm (actual 241 patients per arm), over an estimated period of 24 months. Final analysis would occur at approximately 424 deaths, which was expected to be observed about 43 months after the accrual of the first patient. A stratified log rank analysis would have 90% power to detect a 27.5% reduction in the risk of death, i.e., a hazard ratio of 0.725, between Arm A and Arm C; Test type: Superiority; p < 0.0249, Kaplan-Meier — one-sided; Hazard Ratio (HR) = 1.013, 95% CI 2-sided [0.837 to 1.226]
Statistical Analysis 2: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; Subgroup analyses (pre-specified): Presence of antecedent MDS or MPD (covariate) Treatment covariate: alternating sapacitabine/decitabine treatment Levels: No (i.e., de novo) vs Presence of antecedent MDS or MPD; Test type: Superiority; p < 0.0249, Log Rank — one-sided; Cox Proportional Hazard = 1.08, 95% CI 2-sided [0.86 to 1.35] — Predictive factor adjusted; when interaction term was not significant at 10% confidence level, the interaction term was removed from the model
Statistical Analysis 3: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; Subgroup analyses (pre-specified): Baseline peripheral WBC count ≥ 10 x 109/L (covariate) Treatment covariate: alternating sapacitabine/decitabine treatment Levels: Baseline WBC count ≥ 10 x 109/L vs WBC count ≤ 10 x 109/L; Test type: Superiority — Effects of treatments compared in AML patients with baseline WBC count ≥ 10 x 109/L vs WBC count ≤ 10 x 109/L; p < 0.0249, Log Rank — one-sided; Cox Proportional Hazard = 1.57, 95% CI 2-sided [1.12 to 2.19] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; Subgroup analyses (pre-specified): Baseline bone marrow blast percentage ≥ 50% (covariate) Treatment covariate: alternating sapacitabine/decitabine treatment Levels: Baseline bone marrow blast percentage ≥ 50% vs Blast percentage ≤ 50%; Test type: Superiority; p < 0.0249, Log Rank — one-sided; Cox Proportional Hazard = 1.01, 95% CI 2-sided [0.77 to 1.32] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; Subgroup analyses (pre-specified): Unfavorable cytogenetics risk by SWOG (covariate) Treatment covariate: alternating sapacitabine/decitabine treatment Levels: Unfavorable cytogenetics vs other; Test type: Superiority; p < 0.0249, Log Rank; Cox Proportional Hazard = 1.27, 95% CI 2-sided [0.94 to 1.73] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; Subgroup analyses (post-hoc): Region (covariate) Treatment covariate: alternating sapacitabine/decitabine treatment (Arm A) Levels: EU vs US; Test type: Superiority; p < 0.0249, Log Rank — one-sided; Cox Proportional Hazard = 1.222 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; Subgroup analyses (post-hoc): Age (covariate) Treatment covariate: alternating sapacitabine/decitabine treatment (Arm A) Levels: ≥ 75 years old vs ≤ 75 years old; Test type: Superiority; p < 0.0249, Log Rank — one-sided; Cox Proportional Hazard = 1.071 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; Subgroup analyses (post-hoc): Gender (covariate) Treatment covariate: alternating sapacitabine/decitabine treatment (Arm A) Levels: Male vs Female; Test type: Superiority; p < 0.0249, Log Rank — one-sided; Cox Proportional Hazard = 0.956 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; Subgroup analyses (post-hoc): ECOG status (covariate) Treatment covariate: alternating sapacitabine/decitabine treatment (Arm A) Levels: Status 2 vs < 2; Test type: Superiority; p < 0.0249, Log Rank — one-sided; Predictive factor adjusted; when interaction term was not significant at 10% confidence level, the interaction term was removed from the model
Statistical Analysis 10: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; Subgroup analyses (post-hoc): HCT-CI score (covariate) Treatment covariate: alternating sapacitabine/decitabine treatment Levels: HCT-CI score 0-2 vs HCT-CI score >2; Test type: Superiority; p < 0.0249, Log Rank — one-sided; [statistical method as in outcome 1, analysis 9]

2. Secondary Outcome: Complete Remission (CR)
Description: Normalization of peripheral neutrophils to >=1000 /microliter, platelet to >=100,000/microliter within 2 weeks of bone marrow biopsy/aspirate, and bone marrow to <=5 % blasts; independent of transfusions*; and no extramedullary leukemia.
  * independent of transfusions refer to no platelet transfusion for 1 week prior to achieving the response
Time Frame: up to 43 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 241 | 241
Participants
  Responders | 40 | 26
  Non-Responders | 198 | 213
  Missing | 3 | 2
Statistical Analysis 1: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; Test type: Superiority; p = 0.1468, Fisher Exact; Cox Proportional Hazard = 1.340, 95% CI 2-sided [0.645 to 2.782]

3. Secondary Outcome: Complete Remission With Incomplete Platelet Count Recovery (CRp)
Description: Normalization of bone marrow to <=5% blasts; peripheral neutrophils >=1000 /microliter, platelet <=100,000 /microliter within 2 weeks of bone marrow biopsy/aspirate; independent of transfusions*; and no extramedullary leukemia.
  *independent of transfusions refer to no platelet transfusion for 1 week prior to achieving the response
Time Frame: up to 43 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 241 | 241
Participants
  Responders | 5 | 5
  Non-Responders | 233 | 234
  Missing | 3 | 2

4. Secondary Outcome: Partial Remission (PR)
Description: Normalization of peripheral neutrophils to >=1000 /microliter, platelet to >=100,000/microliter within 2 weeks of bone marrow biopsy/aspirate, >=50% decrease in bone marrow blasts over pre-treatment but still >5%; independent of transfusions*
  *independent of transfusions refer to no platelet transfusion for 1 week prior to achieving the response
Time Frame: up to 43 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 241 | 241
Participants
  Responders | 12 | 8
  Non-Responders | 226 | 231
  Missing | 3 | 2

5. Secondary Outcome: Hematological Improvement
Description: HI with duration (HI)
  1. Erythroid response (HI-E) for patients with pre-treatment hemoglobin < 11 g/dL; Major response: >2 g/dL increase in hemoglobin; for RBC, transfusion independence* Minor response: 1 to 2 g/dL increase in hemoglobin; for RBC, a 50% decrease in transfusion requirements
  2. Platelet response (HI-P) for pre-treatment platelet count <100,000/mm3; Major response: an absolute increase of platelet count by >=30,000/mm3; stabilization of platelet counts and platelet transfusion independence* Minor response: >=50% increase in platelet count with a net increase > 10,000/mm3 but <30,000/mm3
  3. Neutrophil response (HI-N) for absolute neutrophil count (ANC) < 1,500/mm3 before therapy; Major response: >=100% increase, or an absolute increase of >500/mm3, whichever is greater Minor response: >=100% increase, but absolute increase < 500/mm3
     * independent of transfusions refer to no platelet transfusion for 1 week prior to achieving the response
Time Frame: up to 43 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 241 | 241
Participants
  Responders | 41 | 38
  Non-Responders | 197 | 201
  Missing | 3 | 2

6. Secondary Outcome: Stable Disease (SD)
Description: Failure to achieve at least hematologic improvement (HI), but no evidence of clinically significant progression for > 16 weeks.
Time Frame: up to 43 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 241 | 241
Participants
  Responders | 21 | 31
  Non-Responders | 217 | 208
  Missing | 3 | 2

7. Secondary Outcome: Blood Products Transfused
Description: Number of units of packed red blood cells (PRBC) and/or platelet transfusions administered per 8-week period prior to the first dose of study drug and through the date of treatment discontinuation.
Time Frame: up to 43 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Pint
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 236 | 233
Pint | 20 [0 to 337] | 14 [0 to 260]
Statistical Analysis 1: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; Test type: Superiority; p = 0.0416, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Hospitalized Days
Description: In-patient days in hospital.
Time Frame: up to 12 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 236 | 233
Days | 15 [0 to 93] | 14 [0 to 172]
Statistical Analysis 1: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; Test type: Superiority; p = 0.1568, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: 1-year Survival
Description: One-year survival is the percentage of patients who are alive at 1-year measured from the date of randomization.
Time Frame: Percentage of patients alive at 1 year after randomization (participants were assessed up to 43 months for overall survival curve estimation but this measure presents the 1 year survival rate percentage).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 241 | 241
Participants | 81 | 83
Statistical Analysis 1: Comparison: Sapacitabine-decitabine Alternating vs Decitabine; Test type: Superiority; p < 0.0249, Log Rank — one-sided; Cox Proportional Hazard = 1.013, 95% CI 2-sided [0.837 to 1.226]

10. Secondary Outcome: Duration of Complete Remission (dCR)
Description: Durations of normalization of peripheral neutrophils to >=1000 /microliter, platelet to >=100,000/microliter within 2 weeks of bone marrow biopsy/aspirate, and bone marrow to <=5 % blasts; independent of transfusions*; and no extramedullary leukemia.
  * independent of transfusions refer to no platelet transfusion for 1 week prior to achieving the response
Time Frame: up to 43 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 40 | 26
months | 9.5 [6.1 to 13.6] | 10.4 [8.1 to 14.0]

11. Secondary Outcome: Duration of Complete Remission With Incomplete Platelet Count Recovery (dCRp)
Description: Duration of normalization of bone marrow to <=5% blasts; peripheral neutrophils >=1000 /microliter, platelet <=100,000 /microliter within 2 weeks of bone marrow biopsy/aspirate; independent of transfusions*; and no extramedullary leukemia.
  *independent of transfusions refer to no platelet transfusion for 1 week prior to achieving the response
Time Frame: up to 43 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 5 | 5
months | 9.5 [3.1 to 20.7] | 5.7 [3.0 to 12.5]

12. Secondary Outcome: Duration of Partial Remission (dPR)
Description: Duration of normalization of peripheral neutrophils to >=1000 /microliter, platelet to >=100,000/microliter within 2 weeks of bone marrow biopsy/aspirate, >=50% decrease in bone marrow blasts over pre-treatment but still >5%; independent of transfusions*
  *independent of transfusions refer to no platelet transfusion for 1 week prior to achieving the response
Time Frame: up to 43 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 12 | 8
months | 2.2 [1.2 to 9.9] | 1.9 [0.5 to 9.8]

13. Secondary Outcome: Duration of Hematological Improvement (dHI)
Description: Duration of HI
  1. Erythroid response (HI-E) for patients with pre-treatment hemoglobin < 11 g/dL; Major response: >2 g/dL increase in hemoglobin; for RBC, transfusion independence* Minor response: 1 to 2 g/dL increase in hemoglobin; for RBC, a 50% decrease in transfusion requirements
  2. Platelet response (HI-P) for pre-treatment platelet count <100,000/mm3; Major response: an absolute increase of platelet count by >=30,000/mm3; stabilization of platelet counts and platelet transfusion independence* Minor response: >=50% increase in platelet count with a net increase > 10,000/mm3 but <30,000/mm3
  3. Neutrophil response (HI-N) for absolute neutrophil count (ANC) < 1,500/mm3 before therapy; Major response: >=100% increase, or an absolute increase of >500/mm3, whichever is greater Minor response: >=100% increase, but absolute increase < 500/mm3
     * independent of transfusions refer to no platelet transfusion for 1 week prior to achieving the response
Time Frame: up to 43 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 41 | 38
months | 5.8 [2.7 to 17.0] | 4.8 [3.4 to 7.2]

14. Secondary Outcome: Duration of Stable Disease (dSD)
Description: as for outcome 6
Time Frame: up to 43 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sapacitabine-decitabine Alternating | Decitabine
Number analyzed (Participants) | 21 | 31
months | 23.3 [9.1 to 33.2] | 14.8 [10.6 to NA] — Data point not reported in final database. Insufficient number of participants with stable disease.

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the treatment period and in the post-treatment follow-up period (within 28 days after the last dose of study drug if possible or prior to the initiation of new anti-leukemia treatment, whichever comes first) up to 43 months.
Description: The definitions of adverse event and serious adverse event are in congruence with clinicaltrials.gov standard definitions. Note: Other adverse events were not collected for the lead-in phase.
Groups:
- Lead In Phase: Sapacitabine administered in alternating cycles with decitabine
  Sapacitabine: Oral sapacitabine capsules
  Decitabine: Decitabine intravenous
  (n=21, not included in randomization)
Arm/Group | Lead In Phase | Sapacitabine-decitabine Alternating | Decitabine
All-Cause Mortality (participants affected / at risk) | 21/21 | 221/241 | 211/241
Serious Adverse Events (participants affected / at risk) | 17/21 | 199/236 | 188/233
Other Adverse Events (participants affected / at risk) | 0/0 | 236/236 | 232/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead In Phase (N=21) | Sapacitabine-decitabine Alternating (N=236) | Decitabine (N=233)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 51 (478) | 56 (447)
ANAEMIA (Blood and lymphatic system disorders) | 2 (62) | 15 (478) | 14 (447)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 10 (478) | 7 (447)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 7 (478) | 10 (447)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 6 (478) | 3 (447)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (62) | 3 (478) | 6 (447)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (62) | 4 (478) | 5 (447)
DIARRHOEA (Gastrointestinal disorders) | 1 (62) | 5 (478) | 1 (447)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (478) | 5 (447)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 5 (478) | 0 (0)
DISEASE PROGRESSION (General disorders) | 0 (0) | 31 (478) | 19 (447)
PYREXIA (General disorders) | 1 (62) | 10 (478) | 8 (447)
PNEUMONIA (Infections and infestations) | 4 (62) | 56 (478) | 55 (447)
SEPSIS (Infections and infestations) | 1 (62) | 24 (478) | 23 (447)
CELLULITIS (Infections and infestations) | 2 (62) | 10 (478) | 10 (447)
PNEUMONIA FUNGAL (Infections and infestations) | 2 (62) | 4 (478) | 8 (447)
URINARY TRACT INFECTION (Infections and infestations) | 1 (62) | 8 (478) | 4 (447)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 6 (478) | 5 (447)
BACTERAEMIA (Infections and infestations) | 3 (62) | 2 (478) | 6 (447)
INFLUENZA (Infections and infestations) | 0 (0) | 5 (478) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (62) | 2 (478) | 1 (447)
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 (0) | 2 (478) | 1 (447)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (478) | 3 (447)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (62) | 1 (478) | 4 (447)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (447)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (478) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 6 (478) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 3 (478) | 2 (447)
SYNCOPE (Nervous system disorders) | 1 (62) | 3 (478) | 2 (447)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (478) | 3 (447)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 4 (478) | 6 (447)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 2 (478) | 1 (447)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (447)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (478) | 4 (447)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (478) | 5 (447)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (478) | 3 (447)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (478) | 2 (447)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (478) | 2 (447)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (478) | 1 (447)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (478) | 3 (447)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (478) | 3 (447)
HYPERTENSION (Vascular disorders) | 1 (62) | 1 (478) | 1 (447)
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 0 (0) | 1 (478) | 1 (447)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead In Phase (N=0) | Sapacitabine-decitabine Alternating (N=236) | Decitabine (N=233)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | NA | 136 (4020) | 129 (3745)
ANAEMIA (Blood and lymphatic system disorders) | NA | 127 (4020) | 119 (3745)
NEUTROPENIA (Blood and lymphatic system disorders) | NA | 107 (4020) | 88 (447)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | NA | 62 (4020) | 62 (3745)
LEUKOPENIA (Blood and lymphatic system disorders) | NA | 39 (4020) | 27 (3745)
LYMPHOPENIA (Blood and lymphatic system disorders) | NA | 22 (4020) | 19 (3745)
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | NA | 12 (4020) | 12 (3745)
ATRIAL FIBRILLATION (Cardiac disorders) | NA | 23 (4020) | 25 (3745)
SINUS TACHYCARDIA (Cardiac disorders) | NA | 14 (4020) | 20 (3745)
CONSTIPATION (Gastrointestinal disorders) | NA | 85 (4020) | 101 (3745)
NAUSEA (Gastrointestinal disorders) | NA | 98 (4020) | 80 (3745)
DIARRHOEA (Gastrointestinal disorders) | NA | 77 (4020) | 59 (3745)
VOMITING (Gastrointestinal disorders) | NA | 46 (4020) | 39 (3745)
STOMATITIS (Gastrointestinal disorders) | NA | 36 (4020) | 20 (3745)
ABDOMINAL PAIN (Gastrointestinal disorders) | NA | 31 (4020) | 21 (3745)
HAEMORRHOIDS (Gastrointestinal disorders) | NA | 11 (4020) | 17 (3745)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | NA | 9 (4020) | 16 (3745)
FATIGUE (General disorders) | NA | 79 (4020) | 72 (3745)
OEDEMA PERIPHERAL (General disorders) | NA | 72 (4020) | 65 (3745)
PYREXIA (General disorders) | NA | 47 (4020) | 44 (3745)
ASTHENIA (General disorders) | NA | 51 (4020) | 38 (3745)
DISEASE PROGRESSION (General disorders) | NA | 32 (4020) | 20 (3745)
PAIN (General disorders) | NA | 16 (4020) | 14 (3745)
CHILLS (General disorders) | NA | 13 (4020) | 14 (3745)
NON-CARDIAC CHEST PAIN (General disorders) | NA | 8 (4020) | 13 (3745)
PNEUMONIA (Infections and infestations) | NA | 70 (4020) | 69 (3745)
URINARY TRACT INFECTION (Infections and infestations) | NA | 34 (4020) | 22 (3745)
SEPSIS (Infections and infestations) | NA | 27 (4020) | 24 (3745)
CELLULITIS (Infections and infestations) | NA | 17 (4020) | 23 (3745)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | NA | 15 (4020) | 17 (3745)
ORAL CANDIDIASIS (Infections and infestations) | NA | 13 (4020) | 9 (3745)
CONTUSION (Injury, poisoning and procedural complications) | NA | 22 (4020) | 23 (3745)
FALL (Injury, poisoning and procedural complications) | NA | 19 (4020) | 20 (3745)
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | NA | 15 (4020) | 14 (3745)
WEIGHT DECREASED (Investigations) | NA | 53 (4020) | 51 (3745)
BLOOD CREATININE INCREASED (Investigations) | NA | 24 (4020) | 16 (3745)
BLOOD BILIRUBIN INCREASED (Investigations) | NA | 17 (4020) | 22 (3745)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | NA | 11 (4020) | 20 (3745)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | NA | 10 (4020) | 17 (3745)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | NA | 63 (4020) | 54 (3745)
DECREASED APPETITE (Metabolism and nutrition disorders) | NA | 60 (4020) | 51 (3745)
HYPOKALAEMIA (Metabolism and nutrition disorders) | NA | 47 (4020) | 41 (3745)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | NA | 46 (4020) | 41 (3745)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | NA | 35 (4020) | 38 (3745)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | NA | 30 (4020) | 33 (3745)
HYPONATRAEMIA (Metabolism and nutrition disorders) | NA | 15 (4020) | 28 (3745)
DEHYDRATION (Metabolism and nutrition disorders) | NA | 18 (4020) | 18 (3745)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | NA | 14 (4020) | 18 (3745)
FLUID OVERLOAD (Metabolism and nutrition disorders) | NA | 16 (4020) | 13 (3745)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | NA | 38 (4020) | 32 (3745)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | NA | 26 (4020) | 30 (3745)
BACK PAIN (Musculoskeletal and connective tissue disorders) | NA | 27 (4020) | 24 (3745)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | NA | 15 (4020) | 13 (3745)
BONE PAIN (Musculoskeletal and connective tissue disorders) | NA | 10 (4020) | 13 (3745)
HEADACHE (Nervous system disorders) | NA | 39 (4020) | 43 (3745)
DIZZINESS (Nervous system disorders) | NA | 37 (4020) | 31 (3745)
INSOMNIA (Psychiatric disorders) | NA | 29 (4020) | 25 (3745)
ANXIETY (Psychiatric disorders) | NA | 19 (4020) | 19 (3745)
CONFUSIONAL STATE (Psychiatric disorders) | NA | 21 (4020) | 14 (3745)
DEPRESSION (Psychiatric disorders) | NA | 12 (4020) | 17 (3745)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | NA | 15 (4020) | 14 (3745)
DYSURIA (Renal and urinary disorders) | NA | 12 (4020) | 15 (3745)
HAEMATURIA (Renal and urinary disorders) | NA | 8 (4020) | 14 (3745)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | NA | 54 (4020) | 49 (3745)
COUGH (Respiratory, thoracic and mediastinal disorders) | NA | 45 (4020) | 50 (3745)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | NA | 28 (4020) | 29 (3745)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | NA | 21 (4020) | 19 (3745)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | NA | 20 (4020) | 14 (3745)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | NA | 14 (4020) | 10 (3745)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | NA | 12 (4020) | 7 (3745)
RASH (Skin and subcutaneous tissue disorders) | NA | 17 (4020) | 22 (3745)
ALOPECIA (Skin and subcutaneous tissue disorders) | NA | 32 (4020) | 4 (3745)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | NA | 18 (4020) | 17 (3745)
PRURITUS (Skin and subcutaneous tissue disorders) | NA | 15 (4020) | 17 (3745)
PETECHIAE (Skin and subcutaneous tissue disorders) | NA | 17 (4020) | 14 (3745)
ERYTHEMA (Skin and subcutaneous tissue disorders) | NA | 15 (4020) | 13 (3745)
HYPERTENSION (Vascular disorders) | NA | 30 (4020) | 29 (3745)
HYPOTENSION (Vascular disorders) | NA | 18 (4020) | 25 (3745)
HAEMATOMA (Vascular disorders) | NA | 11 (4020) | 10 (3745)

LIMITATIONS AND CAVEATS:
Point to note: The Lead-in AML patients in the sapacitabine-decitabine alternate dosing arm (n=21) were not considered for efficacy assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No